CLINICAL TRIAL: NCT04426903
Title: Application of Cognitive and Physical Training (LLM Care) and Related Affective Computing Systems on People With Parkinson's Disease (Movement Disorders)
Brief Title: Application of LLM Care and Related Affective Computing Systems on People With Parkinson's Disease
Acronym: pdLLM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Panos Bamidis, Professor, Aristotle University Of Thessaloniki
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 490
Record Dates: First submitted 2020-06-09; First posted 2020-06-11 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Parkinson Disease
Keywords: Physical Training; Cognitive Training; EEG; Neuroplasticity
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Participants are assigned to a group following different interventions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LLM Care (Experimental): LLM Care training Participants use the webFitForAll exergaming computer platform as the physical training component (PT); Participants use the language adapted version of the BrainHQ Program as the cognitive training component (CT)
  Interventions: Other: webFitForAll; Other: BrainHQ
- Physical Training (PT) (Experimental): Physical training only. Participants use the webFitForAll exergaming computer platform as the physical training component (PT).
  Interventions: Other: webFitForAll
- Cognitive Training (CT) (Experimental): Cognitive training only. Participants use the language adapted Version of the BrainHQ Program as the cognitive training component (CT).
  Interventions: Other: BrainHQ

INTERVENTIONS:
Other: webFitForAll — PT training participants use the webFitForAll exergaming computer platform as the physical training component (PT)
  Other Names: PT
  Arms: LLM Care; Physical Training (PT)
Other: BrainHQ — CT training participants use the language adapted version of the BrainHQ program as the cognitive training component (CT)
  Other Names: CT
  Arms: Cognitive Training (CT); LLM Care

SUMMARY:
The study is an adaptation of the Long Lasting Memories (LLM) (NCT02267499) and the subsequent LLM Care (NCT02313935) projects in patients with Parkinson's Disease (PD). The study aims to examine the viability and any potential benefits of cognitive and physical training, as offered via the ICT-based (non-pharmacological) intervention of LLM Care, on people with PD. It is worth investigating whether this intervention can offer a better quality of life in patients with PD and counterbalance the often associated with the PD disease neurodegeneration. To evaluate any physical, cognitive, behavioral, and neuroplastic changes and measure the influence (affective status of participant) of the training on the pathological population, the study utilizes somatometric and neuropsychological assessments and neuroscientific (electroencephalographic, EEG-related) indices, as well as affective computing systems.

DETAILED DESCRIPTION:
Parkinson's Disease (PD) is a highly prevalent chronic neurodegenerative disease of the central nervous system, with both motor and non-motor symptoms, having a high impact on the quality of life of the patients. There is still no cure available for individuals with PD but only pharmaceutical treatments that manage the symptoms, thus non-pharmaceutical treatments such as physical and cognitive training are of great importance. This study aims to evaluate the benefits of the LLM Care (NCT02313935) Integrated Healthcare System (https://www.llmcare.gr/en/home/), which is a successful example of commercializing the LLM (NCT02267499) research program (http://www.longlastingmemories.eu/), in patients with PD. The LLM Care (non-pharmaceutical) intervention is an integrated training system that targets nondemented and demented aging population and adopts an approach of cognitive and physical training to improve the quality of life and prolong the functionality of the elders. The physical training (PT) component of the LLM, WebFitForAll, was developed by the research team of the Medical Physics Laboratory, Department of Medicine, Aristotle University of Thessaloniki. WebFitForAll is an effective physical platform that strengthens the body and enhances aerobic capacity, flexibility, and balance. The cognitive training (CT) component of the LLM is a Greek adaptation of the BrainHQ online interactive environment, and comprises six categories with 29 brain exercises with hundred levels of difficulty. The exercises focus on attention, memory, brain speed, people skills, navigation, and intelligence. The target population is PD patients which were classified according to their cognitive state as PD-cognitively normal (PD-CN) and PD-mild cognitive impairment (PD-MCI). Both PD-CN and PD-MCI followed similar training schemes of the intervention, two times per week for one hour for a total of 10 weeks (aiming at 20 sessions/individual). Specifically, the patients were categorized as follows: (i) LLM training group, where participants attended a training protocol consisting of pseudo-randomized physical and cognitive exercises (30 minutes of cognitive and 30 minutes of physical training), (ii) physical training group, whereas participants underwent only physical training (one hour of physical training), and (iii) cognitive training group, in which participants performed cognitive tasks (one hour of cognitive training). The main goal of this study is to quantify the effects of implementing the LLM Care intervention on patients with PD, determine any benefits in physical status, cognition, behavior, and brain function, and eventually assess if adopting a cognitively and physically stimulating lifestyle can offer a better quality of life in this pathological group. All of the patients were evaluated at baseline (pre) and exit (post) via EEG measures and a battery of routinely used clinical and neuropsychological tests. Additionally, the training platform utilizes affective computing systems to evaluate the affective status of all participants throughout the training and to establish a pleasant learning environment for all participants.

ELIGIBILITY:
Inclusion Criteria:

1. Age 50 years and older
2. Native level speakers of the Greek language
3. Able to commit for the required intervention time
4. No significant mobility problems (upper or lower limbs)
5. Normal or corrected to normal visual and auditory acuity
6. In case of any chronic diseases, such as hypertension, diabetes, etc., there should be advice from the competent doctor
7. No serious cardiovascular problems
8. Mild physical activity supervised by a physician
9. Stable medication so as not to affect the patient's functionality from Parkinson's motor symptoms (e.g., stiffness, dyskinesia, restlessness, gait disorder and instability, etc.)

Exclusion Criteria:

1. History of serious neurological diseases or psychiatric illness
2. Recent (within 6 months) history of stroke, transient ischemic stroke episode, traumatic brain injury, ALS, multiple sclerosis
3. Substance abuse
4. Use of acetylcholinesterase inhibitor is not excluded, as long as its use has started 4 months before joining the study, and is stable during its course study remains constant
5. Significant communication disorders
6. Simultaneous enrolment in other studies
7. Patients suspected of not being able or willing to cooperate or comply with study protocol requirements
8. Statin users may be excluded unless during the study the use is constant
9. Patients diagnosed in stages 4 and 5 of the disease, or have undergone surgical treatment

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Change in current density strength of the cortical activity as measured via EEG. | 2 months
  Change is defined as statistical significance in the t-test comparison of the current density strength as reconstructed via Low Resolution Electromagnetic Tomography (LORETA) algorithm on the basis of high-density EEG recordings before compared to after the training.
Changes in the cortical directed connectivity as measured via EEG | 2 months
  Changes in the cortical connectivity caused via the training. Change is defined as statistical significance in the t-test comparison of the Phase Transfer Entropy (PTE) estimated from the cortical activity, as reconstructed via Low Resolution Electromagnetic Tomography (LORETA) algorithm on the basis of high-density EEG recordings, before compared to after the training.
Changes in the graph theory indexes as measured via EEG | 2 months
  Changes in the global and local graph theoretical indexes of the brain networks caused via the training. Change is defined as statistically significance in the t-test comparison of the graph theory indexes, before compared to after the training.

SECONDARY OUTCOMES:
Physical capacity (mobility) | 2 months
  Change in walking speed as measured via the 10 Meter Walk test (Walking Speed m/s; Household Ambulator: <0.40 m/s; Limited Community Ambulator: 0.40 to <0.80 m/s; Community Ambulator: ≥0.80 m/s)
Change in physical capacity (gait and balance, fall risk) | 2 months
  Change in gait and balance, and fall risk as measured via the Tinetti POMA (scale: 0-28; gait is scored over 12; balance is scored over 16; perfect: 28; the lower the score on the Tinetti test, the higher the risk of falling; High risk of fall: ≤ 18; Moderate risk of fall: 19-23; Low risk of fall≥ 24)
Body Weight index | 2 months
  BMI
Fitness | 2 months
  Change in Fitness. Change in aerobic fitness, strength, and flexibility as measured via the Fullerton Senior Fitness Test (SFT)
Physical capacity (balance & mobility) | 2 months
  Community Balance & Mobility: balance and mobility, scale: 0-96 perfect:96
Physical capacity (Functional mobility) | 2 months
  Berg Balance Scale: functional mobility, scale: 0-56 perfect:56
Quality of life index | 2 months
  PDQ-8: activities of daily living, attention and working memory, communication, depression, quality of life, and social relationships in persons with Parkinson's Disease, scale: 0-100 (0: good health, 100: poor health)
Depression | 2 months
  GDS: depressive symptoms, scale: 0-15 (normal: 0-5; mild depression: 5-8; moderate depression: 9-11; severe depression: 12-15)
Physical capacity (general) | 2 months
  Change in physical function as measured via the Short Physical Performance Battery (SPPB, scale from 0 to 12, perfect 12)
Cognitive capacity (functional) | 2 months
  MMSE: orientation, attention, memory, language and visual-spatial skills, scale: 0-30 perfect:30
Cognitive capacity (Visuospatial attention) | 2 months
  Change in visuospatial attention as measured via Trail Making Test (TMT, duration of completion)
Cognitive capacity | 2 months
  Change in cognitive function as measured via the Montreal Cognitive Assessment (MOCA, scale: 0-30; perfect: 30; normal: ≥26)

CONTACTS AND LOCATIONS:
Overall Officials: Panagiotis D bamidis, PhD, Principal Investigator — Professor
Locations (1):
- Laboratory of Medical Physics, AUTH, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Savvidis TP, Konstantinidis EI, Dias SB, Diniz JA, Hadjileontiadis LJ, Bamidis PD. Exergames for Parkinson's Disease Patients: How Participatory Design Led to Technology Adaptation. Stud Health Technol Inform. 2018;251:78-81. PMID 29968606
- [Background] Konstantinidis EI, Bamparopoulos G, Bamidis PD. Moving Real Exergaming Engines on the Web: The webFitForAll Case Study in an Active and Healthy Ageing Living Lab Environment. IEEE J Biomed Health Inform. 2017 May;21(3):859-866. doi: 10.1109/JBHI.2016.2559787. Epub 2016 Apr 27. PMID 28113566
- [Background] Styliadis C, Kartsidis P, Paraskevopoulos E, Ioannides AA, Bamidis PD. Neuroplastic effects of combined computerized physical and cognitive training in elderly individuals at risk for dementia: an eLORETA controlled study on resting states. Neural Plast. 2015;2015:172192. doi: 10.1155/2015/172192. Epub 2015 Apr 7. PMID 25945260
- See also: Related Info — https://www.llmcare.gr/